CLINICAL TRIAL: NCT04287972
Title: A Monocentric Randomized Controlled Prospective Study to Evaluate the Antireflux Efficacy of Primary Crural Closure During Sleeve Gastrectomy for Obese Patients With Incompetents Oeso-gastric Valves
Brief Title: A Study to Reduce the Reflux After a Sleeve Gastrectomy in Obese Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative issues
Sponsor: Fabio Garofalo (Other)
Responsible Party: Sponsor-Investigator, Fabio Garofalo, Sponsor Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORL-CHIR-003
Record Dates: First submitted 2020-01-21; First posted 2020-02-27 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Gastroesophageal Reflux; Obesity
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSG-DPC (Experimental): Laparoscopic Sleeve Gastrectomy and Diaphragmatic Pillar Closure.
  Interventions: Procedure: DPC; Procedure: LSG
- LSG (Active Comparator): Laparoscopic Sleeve Gastrectomy
  Interventions: Procedure: LSG

INTERVENTIONS:
Procedure: DPC — The anterior fat pad is dissected until the left crura is visible, pars flaccida is open and the right crura exposed. Phreno-oesophageal ligament is sectioned starting from the right crura. Posterior and anterior vagal nerve are recognized before the oesophageal dissection. An intra-abdominal oesophagus lengths of 2 or 3 cm is obtained in order to reduce tension. Left and right crura are sutured with 2 or 3 non absorbable 2-0 stitches; an additional anterior stitch is posed if necessary to calibrate hiatus size without oesophageal deviation.
  Arms: LSG-DPC
Procedure: LSG — After omental section close to gastric insertion, gastric stapling is realised with triple line endo stapler (normally 5 or 6 re-loads). The gastrectomy begins 5-6 cm from the pylorus; gastric fundus is totally resected keeping a distance of 5-10 mm from oesophagus. Any bleeding on staple line is controlled with surgical clips or coagulator.

SUMMARY:
This is a monocentric randomized controlled prospective study. A total of 122 patients will be recruited and randomized 1: 1 in the experimental group - Laparoscopic Sleeve Gastrectomy and Diaphragmatic Pillar Closure - or in the control group - Laparoscopic Sleeve Gastrectomy.

At 6 months post surgery a gastroscopy, an oesophageal manometry and a PH-study will be perform to detect de novo GastroEsophageal Reflux Disease and hiatal hernia appearance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Patient with BMI between 35 and 50 Kg/m2 for whom laparoscopic sleeve gastrectomy indication was made
* Patients with no preoperative gastroesophageal reflux disease symptoms
* Hill 2-3 or 4 (with HH <2 cm) hypogastric valve diagnosed preoperatively

Exclusion Criteria:

* Gastroesophageal reflux disease with daily symptoms or daily use of proton pump inhibitors drugs or daily use of anti-H2 drugs
* Hiatal Hernia >2cm and/or esophagitis and/or Barrett metaplasia
* Previous bariatric and/or gastric surgery
* Normal gastroesophageal valve (Hill 1)
* Motility disorders of the esophagus (documented on manometry)
* PH-study positive for gastro-oesophageal reflux disease (DeMeester Score >14.1)
* Contraindications to gastroscopy or manometry or ph-study
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Patient not legally competent
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
De novo GastroEsophageal Reflux Disease (GERD) onset | 6 months post surgery
  At 6 months post surgery a gastroscopy, an oesophageal manometry and a PH-study will be perform to detect de novo GERD (GastroEsophageal Reflux Disease)

SECONDARY OUTCOMES:
hiatal hernia appearance | 6 months post surgery
  At 6 months post surgery a gastroscopy, an oesophageal manometry and a PH-study will be perform to detect hiatal hernia appearance
change in patient-reported quality of life using Gastroparesis Cardinal Symptom Index (GCSI) questionnaire | baseline and 6 months post surgery
  Evaluation of benefits in term of life quality by Gastroparesis Cardinal Symptom Index (GCSI) self-assessment of gastroparesis symptoms.
  The Gastroparesis Cardinal Symptom Index (GCSI), is a questionnaire that assess severity of symptoms associated with gastroparesis. Symptoms are rated from 0 (no symptom) to 5 (very severe)
change in patient-reported quality of life using GERD-Health Related Quality of Life Questionnaire (GERD-HRQL) questionnaire | baseline and 6 months post surgery
  Evaluation of benefits in term of life quality and reduction of Protonic Pomp Inhibitors drugs by GERD-Health Related Quality of Life questionnaire.
  Questionnaire (GERD-HRQL) for symptoms related to GERD. Symptoms are rated from 0 (no symptom) to 5 (Symptoms are incapacitating to do daily activities). The total Score is calculated by summing the individual scores to 15 questions.
  * Greatest possible score (worst symptoms) = 75
  * Lowest possible score (no symptoms) = 0
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months post surgery
  Evaluation of number of participants with treatment-related adverse events ( short and long term surgical complications)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Garofalo, Principal Investigator — EOC
Locations (1):
- Ospedale Regionale di Lugano, Civico e Italiano, Lugano, Switzerland